CLINICAL TRIAL: NCT02118818
Title: Next Generation Sequencing Approach to the Study of Rheumatic Heart Disease
Brief Title: RhEumatiC Heart diseAse Genetics
Acronym: RECHARGE
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National University, Rwanda (Other)
Responsible Party: Principal Investigator, Jochen Daniel Muehlschlegel, MD, Associate Professor of Anesthesia, Brigham and Women's Hospital
Other Study IDs: 2013P002682/BWH
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — The investigators are collecting blood for DNA analysis from all subjects as well as heart valve tissue from subjects who undergo cardiac surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NO rheumatic heart disease by echo: There will be no intervention. This is an observational trial to examine the differences in genetic variants and gene expression between patients with and without RHD. We will be using next generation sequencing to identify these differences.
  Interventions: Genetic: Next generation sequencing
- Rheumatic heart disease by echo: There will be no intervention. This is an observational trial to examine the differences in genetic variants and gene expression between patients with and without RHD. We will be using next generation sequencing to identify these differences.
  Interventions: Genetic: Next generation sequencing

INTERVENTIONS:
Genetic: Next generation sequencing — There will be no intervention. This is an observational trial to examine the differences in genetic variants and gene expression between patients with and without RHD.

SUMMARY:
Rheumatic fever (RF) is an autoimmune disease that is mediated by the cellular and humoral immune response that follows an untreated pharyngeal Streptococcus pyogenes infection. The most serious complication is rheumatic heart disease (RHD), one of the most common problems facing children and young adults worldwide, which leads to chronic valvular lesions. It is estimated that 60% of all acute rheumatic fever cases will develop RHD.

The pathogenesis of RHD is complex with both environmental and genetic factors contributing to its etiology. The investigators know little about the genetic etiology, cellular events and modifiers of progression of RHD, and there exists a wide range of disease severity and progression to severe valve pathology.

Thus, the investigators will study the genetics of RHD in Rwanda, a country with a very high incidence of RHD, using a combination of next-generation targeted exome capture, transcriptomics, and expressed quantitative trait loci (eQTL) analysis.

DETAILED DESCRIPTION:
There are an estimated 2.4 million children between 5 and 14 years of age affected by RF and/or RHD in developing countries of the world, approximately one million of whom live in sub-Saharan Africa (>40%) (1). A systematic review of prevalence studies found exceptionally high rates of RHD in sub-Saharan Africa, with the highest level found at 30.4 cases per 1000 children in Mozambique (2,3,4,5). At present, no specific treatment for rheumatic heart disease exists other than for its complications, including heart failure, atrial fibrillation, ischemic embolic events, and infective endocarditis. Medical treatment (other than antibiotic prophylaxis) has shown little evidence of slowing the progression of the disease. Medical heart failure treatment is given when patients become symptomatic, and includes mainly β blockers, angiotensin converting- enzyme inhibitor therapies, or a combination of both, as tolerated, and symptomatic treatments such as diuretics. Patients with atrial fibrillation need rate or rhythm control and anticoagulation with warfarin if at high risk of embolic complications. Rheumatic heart disease is a major cause of infective endocarditis in African countries.

North American and European guidelines have considerably reduced the number of heart disorders needing antibiotic prophylaxis to prevent infective endocarditis. Whether guidelines issued from developed regions can be safely applied to developing countries is debatable, and further studies are warranted. Pregnancy in patients with rheumatic heart disease is a challenge, and is associated with high morbidity and mortality. Antenatal consultation with support from cardiology and obstetrics clinics should be done to Provide contraception, counseling, treatment planning before start of pregnancy, and planning for patients with moderate to severe disease who are already pregnant (e.g. caesarean section).

Rheumatic fever (RF) is an autoimmune disease that is mediated by the cellular and humoral immune response that follows an untreated pharyngeal Streptococcus pyogenes infection. The most serious complication is rheumatic heart disease (RHD), one of the most common problems facing children and young adults worldwide, which leads to chronic valvular lesions. It is estimated that 60% of all acute rheumatic fever cases will develop RHD. Each year, there are >280,000 new cases and almost as many deaths from RHD, with a worldwide prevalence of >15 million, of which almost 20% are children aged 5-14 years. The worldwide mortality from RHD is 1.5% annually, compared with an overall mortality of 0.26% for all other cardiovascular diseases in the US3. 79% of all RHD cases come from less developed countries with the highest prevalence in sub-Saharan Africa and Pacific and indigenous Australia/New Zealand (~3-7 cases per 1,000).

The pathogenesis of RHD is complex with both environmental and genetic factors contributing to its etiology, though molecular mimicry between components of S. pyogenes and human heart tissue appear to be a central problem. A clear correlation exists between disease prevalence and lower socioeconomic status in developing countries, while the disease prevalence in developed countries continues to decline. However, the manifestation of acute rheumatic fever in only a subset of children with untreated throat infection by S. pyogenes, familial clustering, and high concordance of RHD among monozygous twins provides strong evidence for genetic determinants for disease susceptibility. Yet the investigators know little about the genetic etiology, cellular events and modifiers of progression of RHD, and there exists a wide range of disease severity and progression to severe valve pathology.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and echocardiographic signs of RHD using WHF criteria

Exclusion Criteria:

* Congenital heart disease

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will include patients aged between 5-40 years in Rwanda presenting with an initial diagnosis of RHD and whose echocardiographic findings meet the criteria for definite RHD. World Heart Federation's criteria for echocardiographic diagnosis of definite RHD will be used, utilizing a combination of pathological criteria and morphological features.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2014-02; Primary Completion 2024-07 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Echocardiographic signs of rheumatic heart disease | 3 years
  All patients enrolled will have had an echocardiogram of their heart to assess for signs of rheumatic heart disease according to WHF criteria. The investigators will perform next generation sequencing on their tissue samples and perform a combination of whole exome or genotyping array on their DNA samples. The goal is to identify variants in those patients with severe disease compared to age, gender, socioeconomic, geographically matched controls without echocardiography signs of RHD.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen D Muehlschlegel, MD MMSc, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- University of Rwanda, Kigali, Rwanda